CLINICAL TRIAL: NCT04051216
Title: The SMART CART Study: Health Information Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UMCC 2016.051; HUM00115179 (Other: University of Michigan Rogel Cancer Center)
Record Dates: First submitted 2019-07-25; First posted 2019-08-09 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Leukemia, Acute; Leukemia, Lymphoblastic
Keywords: caregivers; health information technology; patient-centered care
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Fitness Trackers; Interviews as Topic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (Experimental): Caregivers receive the Roadmap information system loaded on an Apple iPad® for use during the inpatient hospitalization of CART therapy. The Roadmap information system consists of 5 modules personalized to the CART patient: laboratory studies, medications, clinical trial enrollment, healthcare providers, and criteria for discharge. Patients wear an activity monitoring device on days 0-100. Patients wear the device as long as they can each day to monitor physical activity level, sleep/wake patterns, skin temperature, heart rate and respiratory rate.
  Interventions: Behavioral: Education information system; Other: Activity monitor; Other: Interview; Other: Survey Administration; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Behavioral: Education information system — Participants will receive a mobile tablet as an educational intervention
  Other Names: Roadmap information system
Other: Activity monitor — Participants will receive at least 1 of 4 activity monitoring devices
Other: Interview — Participants will be interviewed about their experience using the device(s)
Other: Survey Administration — Participants will receive surveys
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This study evaluates the feasibility of using two information technology tools in patients undergoing Chimeric Antigen Receptor T-cell (CART) therapy and other Cytokine Release Syndrome (CRS)-eliciting treatments such as CD123 BITE. The first is an Apple iPad® application called the BMT Roadmap, which shows information about the participant's health. The second is a wearable activity monitoring device. Health information technology tools such as Roadmap system and the activity monitoring device may enable caregivers and patients to become more active participants in their healthcare.

DETAILED DESCRIPTION:
100 patients will be asked to participate in the wearable device portion of the study. 100 caregivers will be asked to participate in the Roadmap (iPad) portion of the study.

Each caregiver will be provided with an iPad to use the BMT Roadmap system. Patients and/or caregivers are free to use this tool as much as they would like on their own time while in the hospital. The hospital care team will collect the iPad when the patient is discharged and ready to go home. Patients and caregivers will also be asked to take three surveys that will ask about their feelings and thoughts about the Roadmap application. The surveys will be completed when patients are admitted for their CART or other CRS-eliciting therapy, when they get discharged from the hospital and around 100 days after they receive their therapy.

In addition to the use of the BMT Roadmap, this study will include around 7-10 interviews about participants' opinions on the two tools and their experience in the therapy process.

ELIGIBILITY:
INCLUSION:

* Caregiver (age 18 years or older) of any patient eligible to undergo therapy in BMT or hematology/oncology that elicits CRS including CART and CD123 BITE and any patient (age 3 years or older) eligible to undergo therapy in BMT or hematology/oncology that elicits CRS including CART and CD123 BITE will be recruited during the "Pre-CART Workup" stage in the outpatient setting.
* CAREGIVER PARTICIPANTS: Caregiver (age 18 years or older) of a patient who will be hospitalized to receive therapy which elicits CRS in the University of Michigan Mott Children's Hospital Adult or Pediatric BMT Units. The age range of patients typically transplanted in the Pediatric BMT unit is 0-25 years, while the Adult BMT unit transplants those older than 25. Caregivers with children (patients) who are younger than 3 years of age may be eligible to participate even though their children are too young to assent or participate themselves.
* PATIENT PARTICIPANTS: Patient (age 10 years or older) who will be hospitalized to receive or after receiving CART therapy will be given the opportunity to assent/consent and participate in the study. With his/her permission, the patient will also be provided with their own iPad® Roadmap information system to use. Qualitative interviews will be conducted in patients (age 10 years or older) with their assent/consent along with neurocognitive testing. Patients (age 10-17.9 years) will be asked to complete surveys that have been validated in this age group and that offer insight into the usefulness of the Roadmap along with neurocognitive testing. Patients (18 years or older) will be asked to complete surveys along with neurocognitive testing. The patient will also be provided with their own non-invasive, wearable activity monitoring device(s) that will track activity and rest levels. Patients 3-9 years old will be enrolled with parental consent but will not be approached for assent. These patients will not be eligible to participate in the survey or interview portions of the study, however, they will be eligible for sample collection, wearable devices and neurocognitive testing.
* Ability to speak and read proficiently in English (the study's instruments have not been translated and validated in languages other than English)
* Willing and able to provide informed consent
* Willing to comply with study procedures and reporting requirements

EXCLUSION:

* Not willing and able to provide informed consent.
* Not willing to comply with study procedures and reporting requirements.

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2017-12-20 (Actual); Primary Completion 2023-08-25 (Actual); Study Completion 2023-11-23 (Actual)

PRIMARY OUTCOMES:
Percentage of caregivers that log onto the BMT Roadmap at least once per day for a minimum of 4 of the 7 days of the week while the patient is in the hospital. | Duration of hospital admission, up to ~6 weeks
  To test the feasibility of implementing the system in the pediatric CART population. This aim will be measured quantitatively by the log-use data.

SECONDARY OUTCOMES:
Percentage of patients who are able to wear the activity monitoring device(s) approximately 12 hours of the day. | Up to day 100 post-CART
  To test the feasibility of implementing a non-invasive, wearable activity monitoring device in the pediatric CART population. This aim will be measured quantitatively by the log-use data.
Percentage of patients from whom longitudinal samples of blood, urine and stool are collected, for correlative studies. | Up to day 100 post-CART
  Feasibility of collecting longitudinal samples of blood, urine and stool from study population. Samples will be used to perform an exploratory analysis of the relationship between these biomarkers and clinical status, Roadmap and wearable device information.
Caregiver activation/participation compared to reference population to measure the impact of Roadmap information system and wearable monitoring device using survey instrument scores of Parent-Patient Activation Measure (P-PAM) as a composite measure. | Up to day 100 post-CART
  Descriptive statistics will be calculated for each Patient Activation Measure (PAM) score and stratified into the appropriate level of activation. Results will be compared with a published sample. Univariate analyses will be performed to assess associations between PAM and demographic, social, and environmental characteristics of the parent (type of insurance, marital status, number of children in household), disease-related characteristics of the patients (age, disease, disease status at CART), satisfaction (Press Ganey, Usefulness), caregiver burden (CQOLC), mood (POMS), anxiety (STAI), stress (Impact of Event Scale-Revised), miscarried helping (HHI), and experiential avoidance (PAAQ). Pearson's correlation (and other suitable measures of association for categorical variables) will be used to determine the nature and significance of association between each variable and Parent-PAM scores. This analysis will not be powered to detect any statistically meaningful differences.
Care providers' satisfaction with the Roadmap information system and non-invasive, wearable activity monitoring device health IT tools for patients and their families/caregivers. | Up to day 100 post-CART
  Qualitative interviews of BMT healthcare providers (physicians, nurses, advanced practitioners, social workers, psychologist, nutritionist, and pharmacologist). This is information gathering only. There is no reference population for this.
Presence of care process redesign associated with the Roadmap information system and wearable monitoring devices. | Up to day 100 post-CART
  Measured qualitatively by semi-structured qualitative interviews.
Quality of care process redesign associated with the Roadmap information system and wearable monitoring devices. | Up to day 100 post-CART
  Measured qualitatively by semi-structured qualitative interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Sung Won Choi, MD, MS, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States